CLINICAL TRIAL: NCT04027842
Title: Effect of 10 Minute-prewarming on Core Body Temperature During Gynecologic Laparoscopic Surgery Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Jin Yong Jung, Professor of anesthesiology and pain medicine, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR-18-174
Record Dates: First submitted 2019-07-12; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Hypothermia; Anesthesia
Keywords: Perioperative hypothermia; Core body temperature; Prewarming; Gynecologic laparoscopic surgery
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prewarming group (Experimental): Participants in Prewarming group was warmed with forced air warming device (WarmTouch WT 6000 Warming Unit, Medtronic, Minneapolis, MN, USA) over the entire body for 10 minutes before anesthesia was induced in the operating theater. All participants received active warming with forced air warming system from the initiation of anesthetic induction until end of surgery.
  Interventions: Device: Prewarming
- Non-prewarming group (No Intervention): In Non-prewarming group, no active warming was conducted before induction of anesthesia. Only standard care was provided with introperative active warming with forced air warming system from the initiation of anesthetic induction until end of surgery.

INTERVENTIONS:
Device: Prewarming — In the operating theater, participants allocated in Prewarming group received 10 min-prewarming, which is cutaneous warming before induction of anesthesia. For prewarming, forced air warming system (WarmTouch WT 6000 Warming Unit, Medtronic, Minneapolis, MN, USA) was used and the warming temperature of the device was set to 45°C.
  Arms: Prewarming group

SUMMARY:
Previous research has shown beneficial effects of prewarming on preventing inadvertent perioperative hypothermia (IPH). Warming the surface of the body before the induction of anesthesia can reduce the temperature difference between the core and periphery, thereby reducing the degree of core-to-peripheral thermal redistribution. It has been proved that initiation of warming before surgery can be more useful for preventing IPH than warming only during surgery. Nevertheless, there are not many researches on effects of short period (<30 min) prewarming, especially in gynecologic laparoscopic surgery. Accordingly, the investigators designed this study to test if IPH can be effectively prevented when 10 minutes of prewarming is added to intraoperative active warming in patients undergoing gynecologic laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 or 2 patients
* patients who underwent gynecologic laparoscopic surgery under general anesthesia

Exclusion Criteria:

* preexisting hypothermia (<36℃) or hyperthermia (>37.5℃)
* anesthesia last for <1 hour or >2 hours
* conversion from laparoscopic surgery to laparotomy
* patients with a body mass index (BMI) ≥ 31kg/m2
* patients with known thyroid disease

Ages: 19 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
the incidence of intraoperative hypothermia | on arrival at operating theater, before anesthesia induced, every 15 minutes after anesthetic induction until admission to the post anesthetic care unit (PACU)
  Number of Participants whose core temperature was than 36℃ was recorded at each time point.

SECONDARY OUTCOMES:
the incidence of postoperative shivering | on the admission to PACU, 30 minutes after the admission to PACU
  Number of Participants who suffer shivering at the post anesthetic care unit was recorded. Postoperative shivering was graded by an investigator who did not know the procedure in the operating room; shivering grade was divided into four grades (0 = none, 1 = mild, 2 = moderate, 3 = severe, The Bedside Shivering Assessment Scale)
Time-temperature interaction during the first 1 hour of anesthesia | Core body temperature was recorded at 15-min intervals from initiation of anesthesia for 1 hour.
  Core body temperature was recorded at each time point. Time-temperature interaction of 2 groups during the first 1 hour of anesthesia was analyzed by RMANOVA

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yong Jung, MD, Principal Investigator — Daegu Catholic University Medical Center
Locations (1):
- DaeguCUMC, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No